CLINICAL TRIAL: NCT05573399
Title: Clinical Efficacy Analysis on Early Oral Feeding Versus Nasojejunal Early Enteral Nutrition for Patients After Pancreaticoduodenectomy
Brief Title: Early Oral Feeding for Patients After Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Guo ShiWei, Research Assistant of Hepatobiliary and Pancreatic Surgery, Changhai Hospital
Other Study IDs: ChanghaiH-PP11
Record Dates: First submitted 2022-10-07; First posted 2022-10-10 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Pancreatoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early oral feeding: No enteral feeding tube was placed after pancreaticoduodenectomy and oral nutrition was given early. Patients were given liquid drinks on the second day after pancreaticoduodenectomy, and solid food from the fifth day.
- Early nasojejunal enteral nutrition: Early enteral nutrition was given early through nasojejunal tube. 5% glucose saline was given on the first day after pancreaticoduodenectomy through nasojejunal tube. Enteral nutrition was given from the second day after pancreaticoduodenectomy. When oral intake was adequate, the nasojejunal tube was removed on the sixth day.

SUMMARY:
This study intends to retrospectively analyze the patients who underwent pancreatoduodenectomy and compare the safety and feasibility between early enteral nutrition through nasojejunal tube and early oral feeding after pancreatoduodenectomy. This study is expected to revise the guidelines for early nutritional support after pancreaticoduodenectomy, reduce postoperative complications, and provide better guidance for clinical work.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy is the standard treatment for periampullary and pancreatic head carcinomas, with the high incidence of perioperative complications ranging from 40% to 60%. Malnutrition is a relevant predictor of post-operative morbidity and mortality after pancreatic surgery. Adequate nutrition is the key to reduce perioperative complications, including abdominal infection, poor healing of wounds, and even gastrointestinal anastomotic leak. The optimal nutritional support method after Pancreaticoduodenectomy is still uncertain, and the current nutritional support methods are diverse. The results of an international survey showed that there was very poor or no agreement on postoperative strategies for the management of nutrition after Pancreaticoduodenectomy. Therefore, the investigators designed this retrospective study to evaluate which was safer and more feasible between early oral feeding and nasojejunal early enteral nutrition after Pancreaticoduodenectomy, using the method of propensity score weighting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent pancreaticoduodenectomy by a certain surgeon in Changhai Hospital
* Patients who were treated with nasojejunal enteral nutrition or oral enteral nutrition after operation.

Exclusion Criteria:

* Patients who underwent pancreaticoduodenectomy by other surgeons during the same period;
* Patients who received other nutritional support rather than nasojejunal tube enteral nutrition or oral enteral nutrition after operation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent pancreaticoduodenectomy in Changhai Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Perioperative complications | From Operation date to three months after operation
  Complications defined by ISGPS in perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, Doctor, Principal Investigator — Changhai Hospital, Shanghai, China
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Jing W, Wu S, Gao S, Shi X, Liu W, Ren Y, Ouyang L, Zheng K, Guo S, Wu C, Jin G. Early oral feeding versus nasojejunal early enteral nutrition in patients following pancreaticoduodenectomy: a propensity score-weighted analysis of 428 consecutive patients. Int J Surg. 2024 Jan 1;110(1):229-237. doi: 10.1097/JS9.0000000000000786. PMID 37755371